CLINICAL TRIAL: NCT04644016
Title: Cord Blood Transplantation in Children and Young Adults With Hematologic Malignancies and Non-malignant Disorders
Brief Title: Cord Blood Transplant in Children and Young Adults With Blood Cancers and Non-malignant Disorders
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-480
Record Dates: First submitted 2020-11-23; First posted 2020-11-25 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: AML; ALL; MDS; MPD Withou Myelofibrosis; NHL or HL; Inherited Metabolic Disorders; Hemoglobinopathies; Bone Marrow Failure; HLH
Keywords: Acute myelogenous leukemia; AML; Myelodysplasia; MDS; Myeloproliferative Disorder; Therapy-Related AML and MDS; Therapy-Related Acute Myeloid Leukemia; T-AML; High-risk cytogenetics; Cord Blood Transplantation; 20-480; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hemoglobinopathies; Bone Marrow Failure Disorders; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts; Myeloproliferative Disorders | interventions — Clofarabine; fludarabine; fludarabine phosphate; Busulfan; Cyclosporins; Mycophenolic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants with malignant hematologic disorders (Experimental): Patients with malignant disorders receive clofarabine intravenously (IV) over 2 hours, fludarabine phosphate (fludarabine) IV over 30 minutes, and busulfan IV over 3 hours on days -5 to -2. Beginning on day -3, patients receive tacrolimus IV or orally (PO) and mycophenolate mofetil IV over at least 2 hours in the absence of unacceptable toxicity. Patients may begin to taper tacrolimus at approximately 3 months post-transplant and mycophenolate mofetil at approximately 60 days post-transplant in the absence of ongoing graft versus host disease (GVHD) requiring systemic immune suppression. TRANSPLANT: Patients undergo cord blood transplantation (CBT) on day 0.**Subgroup will get rATG (day -12 to -10) POST-TRANSPLANT: Beginning on day 7, patients receive filgrastim subcutaneously (SC) or IV over 15-30 minutes until absolute neutrophil count (ANC) recovery. Additionally, patients undergo blood sample collection, computed tomography (CT) and positron emission tomography (PET) on study.
  Interventions: Drug: Clofarabine; Drug: Fludarabine; Drug: Busulfan; Drug: Cyclosporine-A; Drug: Mycophenolate Mofetil; Biological: Cord Blood Graft
- Participants with non-malignant hematologic disorders (Experimental): Patients with non-malignant disorders receive rituximab IV on day -12 and rabbit anti-thymocyte globulin (rATG) over 12 hours on day -12 to -9. Patients then receive clofarabine IV over 2 hours, fludarabine IV over 30 minutes, and busulfan IV over 3 hours on days -5 to -2. Beginning on day -3, patients receive tacrolimus IV or PO and mycophenolate mofetil IV over at least 2 hours. Patients may begin to taper tacrolimus at approximately 6 months post-transplant and mycophenolate mofetil at approximately 60 days post-transplant in the absence of ongoing GVHD requiring systemic immune suppression.
  TRANSPLANT: Patients undergo CBT on day 0. POST-TRANSPLANT: Beginning on day 7, patients receive filgrastim SC or IV over 15-30 minutes until ANC recovery. Patients also receive rituximab IV on day 30.
  Additionally, patients undergo blood sample collection, CT and PET on study.
  Interventions: Drug: Clofarabine; Drug: Fludarabine; Drug: Busulfan; Drug: Cyclosporine-A; Drug: Mycophenolate Mofetil; Biological: Cord Blood Graft

INTERVENTIONS:
Drug: Clofarabine — Clofarabine
  Other Names: Clolar
Drug: Fludarabine — Fludarabine
  Other Names: Fludara
Drug: Busulfan — Busulfan per PK
  Other Names: Busulfex
Drug: Cyclosporine-A — GVHD prophylaxis will consist of cyclosporine-A (CSA) and mycophenolate mofetil (MMF) starting day -3.
  Other Names: CSA
Drug: Mycophenolate Mofetil — GVHD prophylaxis will consist of cyclosporine-A (CSA) and mycophenolate mofetil (MMF) starting day -3.
  Other Names: MMF
Biological: Cord Blood Graft — The CB graft will be infused on day 0 per standard practice
  Other Names: CB graft

SUMMARY:
This is a single-arm study to investigate 1-year treatment related mortality (TRM) in patients with life threatening non-malignant and malignant hematologic disorders who do not have a matched related donor for allogeneic transplantation.

ELIGIBILITY:
Participant Inclusion Criteria:

Age and Donor Status:

Patients with age ≤ 21 years at time of consent with no available and suitably matched related or unrelated donor in the required time period.

Diagnoses :

I. Acute myelogenous leukemia (AML) :

* Complete first remission (CR1) at high risk for relapse such as any of the following:

  * Known prior diagnosis of myelodysplasia (MDS) or myeloproliferative disorder (MPS).
  * Therapy-related AML (t-AML).
  * White cell count at presentation > 100,000.
  * Presence of extramedullary leukemia at diagnosis.
  * Any unfavorable subtype by FAB or WHO classification.
  * High-risk cytogenetics (e.g. those associated with MDS, abnormalities of 5, 7, 8, complex karyotype) or high-risk molecular abnormalities.
  * Requirement for 2 or more inductions to achieve CR1.
  * Presence of Minimal Residual Disease (MRD+) by cytogenetics, flow cytometry or molecular methods after induction.
  * Any patient with newly diagnosed AML with intermediate risk cytogenetics who elects allograft with curative intent over consolidation chemotherapy.
  * Any patient unable to tolerate consolidation chemotherapy as would have been deemed appropriate by the treating physician.
  * Other high-risk features not defined above.
* Complete second remission (CR2).
* Primary refractory or relapsed AML with less than 10% blasts by bone marrow morphology. Patients with cytogenetic, flow cytometric, or molecular abnormalities in ≤ 10% of cells are eligible.

II. Acute lymphoblastic leukemia (ALL):

* Complete first remission (CR1) at high risk for relapse such as any of the following:

  * White cell count at presentation > 30,000 for B-cell lineage and > 100,000 for T-cell lineage.
  * Presence of any high-risk cytogenetic abnormalities such as t (9;22), t (1;19), t (4;11) or other MLL rearrangements (11q23) or other high-risk molecular abnormality.
  * Failure to achieve complete remission (CR) after four weeks of induction therapy.
  * Persistence or recurrence of MRD on therapy.
  * Any patient unable to tolerate consolidation and/or maintenance chemotherapy as would have been deemed appropriate by the treating physician.
  * Other high-risk features not defined above.
* Complete second remission (CR2).
* Primary refractory or relapsed ALL with MRD disease after antibody therapy (e.g., blinatumomab, inotuzumab, other) and/or CAR-T cell therapy.

III. Other acute leukemias:

Leukemias of ambiguous lineage or of other types (e.g. blastic plasmacytoid dendritic cell neoplasm) with less than 5% blasts by BM morphology. Patients with persistent/relapsed disease with cytogenetic, flow cytometric or molecular aberrations in ≤ 5% of cells are eligible.

IV. Myelodysplastic Syndrome (MDS) / Myeloproliferative Disorders (MPD) other than myelofibrosis:

* International prognostic scoring system (IPSS) risk score of INT-2 or high risk at the time of diagnosis.
* Any IPSS risk category if life-threatening cytopenia(s) exists.
* Any IPSS risk category with karyotype or genomic changes that indicate high risk for progression to acute myelogenous leukemia.
* MDS/ myeloproliferative disorder overlap syndromes without myelofibrosis.
* MDS/ MPD patients must have less than 10% bone marrow myeloblasts and ANC ≥ 0.2 (growth factor supported if necessary) at transplant work-up.

V. Non-Hodgkin lymphoma (NHL) or Hodgkin lymphoma (HL) at high-risk of relapse or progression if not in remission:

* Eligible patients with aggressive histology (such as, but not limited to, diffuse large B-cell NHL, mantle cell NHL, and T-cell histology) in CR.
* Eligible patients with indolent B cell NHL (such as, but not limited to, follicular, small cell or marginal zone NHL) will have 2nd or subsequent progression with stable disease/ CR/ PR with no single lesion equal to or more than 5 cm.
* Eligible patients with HL will be those without progression of disease (POD) after salvage chemotherapy with no single lesion ≥ 5 cm.

VI. Inherited Metabolic Disorders [also see EBMT Handbook for discussion on patient eligibility for allogeneic transplant; in general, patients are considered early in the disease course, before they develop neurologic symptoms (46)]:

* Hurler Syndrome
* Hunter (MPS 2 - early disease)
* Sly syndrome (MPSVIII)
* α-Mannosidosis
* X- ALD
* Osteopetrosis
* Metachromatic Leukodystrophy
* Globoid (GLD)

VII. Non-Malignant disorders (other) [also see EBMT Handbook for criteria for transplant (46)]

* Hemoglobinopathies
* Bone Marrow Failure syndromes
* Immunodeficiencies, including HLH

Organ Function and Performance Status Criteria:

* Karnofsky or Lansky score ≥ 70% (see Appendix)
* Bilirubin ≤ 1.5 mg/dL (unless benign congenital hyperbilirubinemia).
* ALT ≤ 3 x upper limit of normal.
* Pulmonary function (spirometry and corrected DLCO) ≥ 50% predicted (corrected for hemoglobin) .
* Left ventricular ejection fraction ≥ 50%.
* Age-adjusted Hematopoietic Cell Transplantation-Comorbidity Index (aaHCT-CI) less than or equal to 7.
* Renal: serum creatinine ≤ 1.5x normal for age. If serum creatinine is outside the normal range, then CrCl > 50 mL/min/1.73m2 (calculated or estimated) or GFR (mL/min/1.72m2) >30% of predicted normal for age.

Normal GFR in Children and Young Adults (Age) : Mean GFR +- SD (mL/min/1.73 m2)

1 week: 40.6 + / - 14.8 2-8 weeks: 65.8 + / - 24.8 >8 weeks: 95.7 + / - 21.7 2-12 years: 133.0 + / - 27.0 13-21 years (males): 140.0 + / - 30.0 13-21 years (females: 126.0 + / - 22.0

GFR, glomerular filtration rate; SD, standard deviation greater than 2 years old: Normal GFR is 100 mL/ min. Infants: GFR must be corrected for body surf ace area.

For metabolic diseases: disease status to be evaluated according to EBMT Handbook [45].

Graft Criteria

CB units will be selected according to the current MSKCC unit selection algorithm. High resolution 8 allele HLA typing and recipient HLA antibody profile will be performed. Cord unit selection will occur based on HLA-match, total nucleated cell (TNC) and CD34+ cell dose adjusted per patient body weight. The cord bank of origin will also be considered. Donor specific HLA antibodies, if present, will also be taken into consideration and may influence the selection of the graft. CB graft will consist of one or two CB units (CBU) based on MSKCC selection algorithm.

* Each CB unit must be at least 3/8 HLA-matched to the patient considering high-resolution 8-allele HLA typing.
* For malignant diseases follow MSKCC CBU selection algorithm
* For non-malignant diseases, CBU will be required to have > 5 x 107 TNC/kg; high HLA allele level match is preferable

Participant Exclusion Criteria:

* Inadequate performance status/ organ function.
* Advanced metabolic disease (EBMT handbook).
* Active CNS leukemic involvement.
* Indolent NHL or Hodgkin lymphoma with progression of disease after most recent salvage chemotherapy.
* Diagnosis of myelofibrosis or other malignancy with moderate-severe bone marrow fibrosis.
* Autologous stem cell transplant within the preceding 6 months.
* Any prior allogeneic stem cell transplant.
* Active and uncontrolled infection (bacterial/fungal/viral) at time of transplantation.
* HIV infection.
* Seropositivity for HTLV-1.
* Pregnancy or breast feeding.
* Patient or guardian unable to give informed consent or unable to comply with the treatment protocol including appropriate supportive care, long-term follow-up, and research tests.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Treatment related mortality at 1 year after myeloablative cord transplant | 1 year
  The primary objective of this study is to assess treatment related mortality (TRM) at 1 year after myeloablative cord transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cancio, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org